CLINICAL TRIAL: NCT05470283
Title: Phase I, Open-Label, Study of Tumor Infiltrating Lymphocytes Engineered With Membrane Bound IL15 Plus Acetazolamide in Adult Patients With Metastatic Melanoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0356; NCI-2022-06873 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2022-07-20; First posted 2022-07-22 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Tumor; Metastatic Melanoma; Melanoma
MeSH Terms: conditions — Neoplasms; Melanoma | interventions — Acetazolamide; Cyclophosphamide; Furosemide; Mesna; fludarabine phosphate; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- OBX-115 plus Acetazolamide (Experimental): Participants will receive chemotherapy to prepare your body for the study drug combination, then you will receive OBX-115 and acetazolamide.
  Interventions: Drug: OBX-115; Drug: Acetazolamide; Drug: Cyclophosphamide; Drug: Furosemide; Drug: Mesna; Drug: Fludarabine Phosphate

INTERVENTIONS:
Drug: OBX-115 — Given by IV
Drug: Acetazolamide — Given by PO
Drug: Cyclophosphamide — Given by IV
  Other Names: Cytoxan®; Neosar
Drug: Furosemide — Given by IV
Drug: Mesna — Given by IV
Drug: Fludarabine Phosphate — Given by IV
  Other Names: Fludarabine; Fludara

SUMMARY:
The goal of this clinical research study is to find the recommended dose of OBX-115 in combination with acetazolamide that can be given to patients with metastatic melanoma previously treated with immune checkpoint inhibitors. The safety and tolerability of the study drug combination will also be studied.

DETAILED DESCRIPTION:
Primary Objective:

• Assess the safety and tolerability of OBX-115 + acetazolamide by CTCAE version 5 criteria to provide a recommended Phase II dose

Secondary Objectives:

* Assess preliminary efficacy of OBX-115 + acetazolamide cell therapy in patients with immune checkpoint inhibitor (ICI)-relapsed and/or refractory metastatic melanoma by evaluating overall response rate (ORR; complete response [CR] + partial response [PR]) by RECIST 1.1 criteria
* Evaluate feasibility of the manufacturing process
* Evaluate duration of response (DOR)
* Evaluate progression free survival (PFS)
* Characterize in vivo cellular kinetics of OBX-115 cells in tumor and/or in peripheral blood by polymerase chain (PCR) and/or fluorescence-activated cell sorting (FACS) analyses
* Characterize the pharmacokinetic profile of acetazolamide when administered in combination with OBX-115
* Characterize the incidence and prevalence of OBX-115 therapy immunogenicity

Exploratory Objectives:

* Assess relationship of soluble immune factors and pharmacodynamic markers, with cellular kinetics, safety, and efficacy
* Describe the composition of OBX-115 subsets (immunophenotyping in peripheral blood mononuclear cells [PBMCs] and in tumor), summarized by clinical response
* Explore the correlation of OBX-115 kinetics in tumor and peripheral blood with clinical endpoints
* Explore the correlation of immune checkpoints with OBX-115 cellular kinetics and efficacy
* Evaluate overall survival (OS)

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients age ≥ 18 at the time of signing ICF
2. Patient has a pathologically confirmed diagnosis of metastatic melanoma that is unresectable stage III or stage IV and has lesion(s) amenable to resection for the generation of TILs and at least one separate lesion for RECIST v1.1 response assessment
3. Patient must be relapsed and/or refractory to immune checkpoint inhibitor (ICI) therapy including either anti PD-1 either with or without anti CTLA-4 blocking antibody and/or anti LAG-3 antibody. Patients should have received standard-of-care (SOC) therapy per standard clinical practice guidelines. Patients must not have had exposure to more than 3 prior lines of anti-PD-1 antibody-containing therapeutic regimens administered in the metastatic setting If the patient is BRAF V600 mutation-positive with rapidly progressing disease, the patient should have received available FDA-approved targeted therapy.
4. ECOG Performance status 0-1
5. Within 7 days of tumor harvest and within 7 days of initiating lymphodepletion, patients must meet the following laboratory criteria:

   • Absolute neutrophil count (ANC) ≥ 1000/mm3

   • Hemoglobin ≥ 8.0 g/dL (transfusion allowed)

   • Platelet count ≥ 75,000/mm3

   • ALT/SGPT and AST/SGOT ≤ 2.5 x the upper limit of normal (ULN)

   • Patients with liver metastases may have liver function tests (LFT) ≤ 5.0 x ULN

   • Calculated creatinine clearance (Cockcroft-Gault) ≥ 50.0 mL/min

   • Total bilirubin ≤ 1.5 X ULN

   • Negative serum pregnancy test (female patients of childbearing potential)
6. Patients must have a 12-lead electrocardiogram (EKG) showing no active ischemia and Fridericia's corrected QT interval (QTcF) less than 480 ms
7. Patients must have echocardiogram showing no evidence of congestive heart failure (as defined by New York Heart Association Functional Classification III or IV) or LVEF <50%
8. Women of child-bearing potential (WCBP), defined as a sexually mature woman who has not undergone a hysterectomy or tubal ligation or who has not been naturally postmenopausal for at least 24 consecutive months, must have a negative serum pregnancy test prior to treatment. All sexually active WCBP and all sexually active male patients must agree to use effective methods of birth control throughout the study. Approved methods of birth control are as follows:

   • Hormonal contraception (i.e. birth control pills, injection, implant, transdermal patch, vaginal ring),

   • Intrauterine device (IUD),

   • Tubal Ligation or hysterectomy,

   • Subject/partner status post vasectomy,
   * Implantable or injectable contraceptives, and
   * Condoms plus spermicide.
9. Patient (or legally authorized representative) has voluntarily agreed to participate in the study by providing signed and dated informed consent (ICF) in accordance with International Conference on Harmonization (ICH) Good Clinical Practice (GCP) guidelines and applicable local regulations
10. Patient has agreed to abide by all protocol required procedures including study related assessments, and management by treating institution for the duration of the study and long-term follow-up (LTFU)
11. Patients who have received bridging therapy between time of TIL harvest and initiation of lymphodepletion must meet all required clinical, laboratory and imaging criteria in order to qualify for therapy initiation
12. Lesions amenable to radiotherapy or palliative radiotherapy (e.g.- bone metastases or metastases causing nerve impingement) should be treated > 4 weeks prior to enrollment and subjects must be fully recovered from the effects of radiation. However, palliative radiation is permitted if subjects recover from all side effects to ≤ Grade 1 toxicities (based on CTCAE, v.5) and is > 2 weeks prior to starting lymphodepletion.

Exclusion Criteria:

1. Patients with uncontrolled intercurrent medical illnesses, including active systemic infection, coagulation disorders or major cardiovascular, respiratory or immune diseases. PI or his/her designee shall make the final determination regarding appropriateness of enrollment
2. Patients on chronic steroid therapy for primary immunodeficiency; however, prednisone or its equivalent is allowed at ≤ 10 mg/day
3. Patients who are pregnant or breastfeeding
4. Chemotherapy within 2 weeks prior to TIL harvest
5. Treatment with small molecule targeted antineoplastics and chemotherapy within 2 weeks of initiation of lymphodepletion, or 5 half-lives, whichever is shorter
6. The use of immune checkpoint inhibitors as bridging therapy is not allowed.
7. Patients who have received live vaccines within 30 days prior to TIL harvest and initiation of lymphodepletion
8. Patients with active infection requiring systemic therapy or causing fever (temperature > 38.1oC) or patients with unexplained fever (temperature > 38.1oC) within 7 days prior to day of investigational product administration
9. Patient has active infection with human immunodeficiency virus (HIV), hepatitis B virus, hepatitis C virus (HCV) requiring active antiviral therapy.
10. Cytomegalovirus (CMV) IgM antibody titer or PCR assay; and Epstein-Barr virus (EBV) IgM or PCR assay indicating active infection. Tumor harvest may take place even with positive results as long as consult with infectious disease physician is planned and the infection can be appropriately treated, if needed, prior to initiation of lymphodepletion.
11. Positive herpes simplex virus (HSV)-1 serology or PCR assay • Patients who are HSV PCR assay positive will need to receive appropriate treatment and become PCR assay negative prior to starting the lymphodepletion Tumor harvest may take place even with positive results as long as consult with infectious disease physician is planned and the infection can be appropriately treated, if needed, prior to initiation of lymphodepletion.
12. Persistent prior therapy-related toxicities greater than Grade 2 according to Common Toxicity Criteria for Adverse Events (CTCAE) v5.0, except for peripheral neuropathy, alopecia, or vitiligo prior to enrollment. Patients with prior immune mediated hypophysitis or adrenal insufficiency or hypothyroidism are eligible for treatment as long as they are on stable, physiologic doses of hormone repletion.
13. History of organ or hematopoietic stem cell transplant
14. History of clinically significant autoimmune disease

The following are exceptions to the criterion:

1. Patients with vitiligo or alopecia.
2. Patients with hypothyroidism, type 1 diabetes or adrenal insufficiency stable on hormone replacement therapy.
3. Patients without active disease in the last 5 years may be included but only after consultation with the PI.
4. Any other history or questionable history of autoimmune disease is to be considered after consultation with the PI

15. History of central nervous system metastases and/or leptomeningeal spread of melanoma.

16. Patients with significant clinical cardiac abnormalities:

• Left ventricular ejection fraction (LVEF) <50%

• congestive heart failure, defined by New York Heart Association Functional Classification III or IV

• unstable angina

* serious uncontrolled cardiac arrhythmia
* a myocardial infarction within 6 months prior to study entry or a history of myocarditis

  17. Patients with a history of interstitial lung disease

  18. History of a concurrent second malignancy (diagnosed in the last 2 years). Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, localized thyroid cancer or in situ cervical cancer that has undergone potentially curative therapy.

  19. Patients unable to provide informed consent and follow the study procedures (e.g., due to language problems, psychological disorders, dementia).

  20. Documented severe/life threatening sulfa allergy.

  21. Chronic need for acetazolamide or other carbonic anhydrase inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-09-07 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Incidence and nature of dose-limiting toxicities (DLTs) during the first 28 days after OBX-115 + acetazolamide administration as assessed by CTCAE version 5.0. Incidence and severity of AEs and SAEs after OBX-115 + acetazolamide administration. | through completion of study, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Rodabe N Amaria, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org